CLINICAL TRIAL: NCT03146767
Title: The Staircase Phenomenon and His Implications on Neuromuscular Block Monitoring During General Anesthesia
Brief Title: The Staircase Phenomenon Implications on Neuromuscular Block Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Anesthesiology Consultant, Hospital Universitario La Fe
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MAZ0816
Record Dates: First submitted 2017-04-25; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Neuromuscular Blockade Monitoring

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No

ARMS (2):
- Tetanic Group (Experimental): A Tetanic stimulation (Tetanus stabilization of baseline) is administered to the monitorized arm before calibrating the neuromuscular block monitor. Then Train-of-four (TOF) stimuli are administered every 20 seconds for 20 minutes.
  Interventions: Device: Tetanus stabilization of baseline
- Control Group (No Intervention): Conventional monitor baseline stabilization: Train-of-four stimuli are administered every 20 seconds for 20 minutes

INTERVENTIONS:
Device: Tetanus stabilization of baseline — Administering a Tetanic stimulus before baseline stabilization shortens the stabilization period of baseline of a neuromuscular block monitor. This acts on the baseline value
  Arms: Tetanic Group

SUMMARY:
The staircase phenomenon could have repercussions on the onset and recovery time following administration of a neuromuscular blocking agent. The investigators aim to assess the magnitude of the staircase phenomenon and its impact on various aspects of neuromuscular blockade with a randomized controlled double blind trial.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiology surgical risk scale) grade I - II
* Surgery not involving airway performed under general anaesthesia with neuromuscular blocker

Exclusion Criteria:

* Pregnancy
* BMI (Body Mass Idex) > 35 Kg/m2
* Anticipated difficult airway
* Chronic kidney or hepatic failure
* Neuromuscular disease
* Medication that has known interactions with neuromuscular blockers
* Hemodynamic failure
* Anticipated large blood loss

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Difference in Block Onset time difference (seconds) | rom 0 seconds up to 240 seconds after neuromuscular block administration at the beginning of surgery. Time frame is the duration of general anesthesia before, during and after surgery (up to 4 hours).
  Onset time is the time between Train of Four (TOF) at the moment of injection of neuromuscular blocking drug and the minimum value reached (onset of neuromuscular block)

SECONDARY OUTCOMES:
Difference in time until recovery of a TOF ratio (TOFr) of 0.9 | From administration of neuromuscular blocking drug until spontaneous reversal (up to 4 hours). Time frame is the duration of general anesthesia before, during and after surgery (up to 4 hours).
  Time until recovery of a TOF ratio of 0.9 (reversal of neuromuscular block as assessed by the monitor). During recovery phase stimuli regain height until all four stimuli of the Train-of-Four are present. Train-of-Four ratio is the ratio between the fourth and the first stimuli (T4/T1).
Difference in TOFr 0.9 Normalized | From administration of neuromuscular blocking drug until spontaneous reversal at this specified point (up to 4 hours). Time frame is the duration of general anesthesia before, during and after surgery (up to 4 hours).
  Time until recovery of a TOF ratio of 0.9 normalized to baseline TOR ratio after calibration. (e.g. if baseline TOF ratio is 1.1, normalized TOF ratio 0.9 is: 1.1 x 0.9 = 0.99)
Difference in time until recovery of 25% of maximum twitch height ot T1 stimulus (DUR25) | From administration of neuromuscular blocking drug until spontaneous reversal at this specified point (up to 4 hours). Time frame is the duration of general anesthesia before, during and after surgery.(up to 4 hours)
  Difference in time until recovery of 25% of maximum twitch height ot T1 stimulus during recovery phase. During recovery phase stimuli begin to recover and their height increases. This outcome is the time between the beginning of neuromuscular block until recovery of 25% of height of the first stimulus of the Train-of-Four.recovery phase. During recovery phase stimuli begin to recover and their height increases. This outcome is the time between the beginning of neuromuscular block until recovery of 25% of height of the first stimulus of the Train-of-Four (TOF)
Time between 25% and 75% of maximum twitch height recovery of T1 stimulus | From administration of neuromuscular blocking drug until spontaneous reversal (up to 4 hours). Time frame is the duration of general anesthesia before, during and after surgery (up to 4 hours).
  Time between 25% and 75% height recovery of maximum twitch height in the recovery phase.
Difference between first stimulus of Train-of-Four ratio at baseline | Single measurement of muscle response after calibration procedure at the beginning of data recording after randomization. It is not a time-to-event variable
  Difference between T1 at baseline. Train-of-Four ratio is the administration of four consecutive stimuli to the monitored muscle. These stimuli are named T1,T2,T3,T4. This is the difference between tow arms oh T1 height at baseline
Difference between T1 height after stabilization period of 20 minutes | Single measurement after 20 minutes stabilization period after beginning of neuromuscular stimulation. It is not a time-to-event variable
  Difference between T1 height after stabilization period of 20 minutes
Difference between TOF ratio at baseline time | Single measurement of muscle response after calibration procedure at the beginning of data recording.
  Difference between TOF ratio at baseline time
Difference between TOF ratio after stabilization period time | Single measurement after 20 minutes stabilization period after beginning of neuromuscular stimulation.
  Difference between TOF ratio after stabilization period time
Monitor Sensitivity difference between groups | Single value no time frame. Sensitivity is internally set by the monitor during calibration (at the beginning of data recording after randomization)
  Sensitivity parameter is set by monitor after calibration.
Monitor Amperage Intensity after calibration difference (milliAmperes, mA) | Single value no time frame. Sensitivity is internally set by the monitor during calibration (at the beginning of data recording after randomization)
  Monitor Amperage Intensity is set by the monitor after calibration
T1/TOFratio relationship difference | Ratio of specified values recorded by the monitor at the beginning of surgery until onset of neuromuscular block (up to 180 seconds) and during spontaneous recovery up to 4 hours until end of anesthesia
  During recovery phase T1 over TOF ratio will be calculated and the difference between two groups will be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario La Fe, Valencia, Spain